CLINICAL TRIAL: NCT06725017
Title: A Phase 2, Multi-center, Randomized, Double-blind, Placebo-Controlled Study to Evaluate the Efficacy and Safety of Live SK08 Powder (Bacteroides Fragilis) in Adult Patients with Active Mild to Moderate Ulcerative Colitis
Brief Title: A Phase 2 Study to Evaluate the Efficacy and Safety of Live SK08 Powder in Adult Patients with Active Mild to Moderate Ulcerative Colitis
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Guangzhou Zhiyi Biotechnology Co., Ltd. (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: SK08UC-201
Record Dates: First submitted 2024-12-05; First posted 2024-12-09 (Actual); Last update posted 2024-12-16 (Actual); Status verified 2024-12

CONDITIONS: Ulcerative Colitis (UC)
Keywords: Ulcerative Colitis
MeSH Terms: conditions — Colitis, Ulcerative

STUDY DESIGN:
Intervention Model Description: randomized, double-blind, placebo-controlled
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (3):
- SK08 low dose group (Experimental): 1 × 10^7 CFU ~ 2.5 × 10^8 CFU/dose, twice daily (BID), taken orally for 8 weeks
  Interventions: Drug: Live SK08 powder
- SK08 high dose group (Experimental): 1 × 10^9 CFU ~ 2.5 × 10^10 CFU/dose, BID, taken orally for 8 weeks
  Interventions: Drug: Live SK08 powder
- Placebo group (Placebo Comparator): BID, taken orally for 8 weeks.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Live SK08 powder — SK08 is an investigational live biotherapeutic product containing a nontoxigenic B. fragilis(NTBF) strain as an active ingredient.
  Arms: SK08 high dose group; SK08 low dose group
Drug: Placebo — Placebo
  Arms: Placebo group

SUMMARY:
This is a Phase 2, multi-center, randomized, double-blind, placebo-controlled study to preliminarily evaluate the efficacy and safety of SK08 in adult patients with active mild to moderate UC. Each subject will undergo three study periods: screening, induction treatment period and a safety follow-up period.

ELIGIBILITY:
Inclusion Criteria:

1. Subjects who voluntarily sign the informed consent form and are able to comply with the study protocol and have the ability to follow relevant procedures.
2. Male and female subjects aged 18-75 years (inclusive) at the time of signing the informed consent.
3. Ulcerative colitis diagnosed by routine clinical, endoscopy, and pathologic criteria for at least 3 months.
4. Subjects with active mild to moderate UC as defined by modified Mayo Score (mMS) of 4-10 (both inclusive), including an endoscopy sub-score of at least 2 and a rectal bleeding sub-score of at least 1.
5. The lesion extends beyond the rectum (colonoscopy shows that the lesion is > 15 cm from the anal verge).
6. Have had no response to, an inadequate response to, or an intolerance to standard 5-ASA treatment (including 5-ASA local treatment), no response or inadequate response means patients have persistent symptoms during treatment with 5-ASA at the recommended dose and treatment duration, intolerance means patients discontinue the 5-ASA treatment due to adverse events. Subjects receiving concurrent stable dose 5-ASA (i.e. no change in medication within 4 weeks of study enrollment and is not expected to change during the study) are permitted to be enrolled.
7. If female, the subject is non-lactating, and is either: Not of childbearing potential, defined as postmenopausal for at least 1 year or surgically sterile due to bilateral tubal ligation, bilateral oophorectomy, or hysterectomy; Of childbearing potential and is practicing at least 1 highly effective method of birth control including the barrier method; oral or parenteral contraceptives; a vasectomized partner; or abstinence from sexual intercourse from the time of signing informed consent and until at least 3 months after the last dose of the study drug. The Investigator will discuss with the subject the option of practicing more than 1 of the above methods for the duration of the study. Subjects must have a negative serum pregnancy test within 7 days prior to the first dose of the study drug.
8. If male and partner is of childbearing potential, the subject agrees to practice at least one highly effective method of birth control from the time of signing the informed consent until at least 3 months after the last dose of the study drug.

Exclusion Criteria:

1. Subjects with Crohn's disease, radiation colitis, diverticulitis, ischemic colitis, microscopic colitis, drug-related (e.g., NSAIDs, tretinoin, immune checkpoint inhibitors, mycophenolate, etc.) colitis, patients with indeterminate colitis, and patients with endoscopy/biopsy showing ileitis/granulomas with clinical suspicion of Crohn's disease.
2. Malignancy or history of malignancy within the previous 5 years except for resected cutaneous basal cell or squamous cell carcinoma that has been treated with no evidence of recurrence.
3. Subjects who received surgery within 30 days before the first dose of study drug or who plan to undergo surgery during the study.
4. Subjects with other pathological conditions in the intestine, including colon dysplasia, intestinal stricture, tumor, intestinal fistula, intestinal obstruction, celiac disease, etc.
5. Presence of any active or chronic recurrent infections.
6. Subjects with previous colectomy, ostomy, J-pouch, or previous intestinal surgery (excluding cholecystectomy, appendectomy).
7. Subjects with severe, progressive or uncontrolled renal, hepatic, hematological, endocrine, immune, cardiovascular, respiratory, neurological, or psychiatric disease.
8. Subjects with poor concurrent medical risks with a clinically significant co-morbid disease such that, in the opinion of the Investigator, the subject should not be enrolled including: Subjects with decompensated liver cirrhosis (Child-Pugh Class B or C) or uncontrolled liver disease; History of pancreatitis; QTc > 450 msec or QTc > 480 msec for participants with bundle branch block at screening and Day 1. The QTc is the QT interval corrected for heart rate according to Fridericia's formula (QTcF); Prior history of bone marrow transplant; Known Hypogammaglobulinemia; Known severe immunodeficiency; AST ≥ 2 × the upper limit of normal (ULN) and/or ALT ≥ 2 × ULN and/or total bilirubin ≥ 2 × ULN; eGFR < 60 mL/min/1.73 m² by Chronic Kidney Disease Epidemiology Collaboration equation (CKD-EPI) calculation; Absolute neutrophil count (ANC) < 500 cells/μL.
9. Subjects with anti-hepatitis C virus (HCV) antibody positive, human immunodeficiency virus (HIV) antibody positive, or hepatitis B surface antigen (HBsAg) positive and need antiviral therapy during the screening period.
10. Subjects have known or suspected hypersensitivity to the study drug and its excipients (maltodextrin, silicon dioxide, magnesium stearate).
11. Subjects who cannot discontinue steroid hormones (such as budesonide multi-matrix (MMX)) oral/topical (suppositories, enemas, etc.), or systemic corticosteroids within 2 weeks before the first dose of study drug.
12. Patients who cannot discontinue other drugs that affect gastrointestinal function, including systemic antibiotics, anti-diarrheal agents, etc., within 2 weeks before the first dose of study drug.
13. Received any probiotic medicines or fecal bacteria transplant within 30 days prior to the first dose.
14. Received treatment with biological agents (infliximab, adalimumab, golimumab, certolizumab, vedolizumab, ustekinumab, natalizumab, etc.) within 8 weeks before the first dose (or 5 half lives of the drug); or received any non-biological agents (cyclosporine, tacrolimus, thalidomide, methotrexate, tofacitinib, etc.) treatment within 30 days before the first dose (or 5 half-lives of the drug).
15. Received (attenuated) live vaccination within 4 weeks of Day 1 or plan to receive during the study until follow-up.
16. Subjects who have participated in any clinical trial within 3 months before screening.
17. Subjects with a history of alcohol and drug abuse.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2025-07-01 (Estimated); Primary Completion 2027-07-01 (Estimated); Study Completion 2027-08-01 (Estimated)

PRIMARY OUTCOMES:
Proportion of subjects achieving clinical remission at Week 8 | 0-8 weeks
  Clinical remission is defined as a total mMS score of 0 to 2, including the following three components:
  * Stool frequency sub-score = 0 or 1.
  * Rectal bleeding sub-score = 0
  * Centrally read endoscopy sub-score = 0 or 1 (score of 1 modified to exclude friability)

SECONDARY OUTCOMES:
proportion of subjects with clinical response at Week 8 | 0-8 weeks
  Clinical response is defined as a decrease from baseline in the total mMS of ≥ 2 points and at least a 30 percent reduction from baseline, and a decrease in rectal bleeding subs-core of greater than or equal to 1 or an absolute rectal bleeding sub-score of 0 or 1.
proportion of subjects with endoscopic improvement at Week 8 | 0-8 weeks
  Endoscopic improvement is defined as a centrally read endoscopy sub-score of 0 or 1.
proportion of subjects with endoscopic remission at Week 8 | 0-8 weeks
  Endoscopic remission is defined as a centrally read endoscopy sub-score of 0.
change from baseline in the total modified Mayo Score at Week 8 | 0-8 weeks
mean change in rectal bleeding and stool frequency sub-scores from baseline to Weeks 2, 4, 6 and 8 | 0-2, 0-4, 0-6, 0-8 weeks

OTHER OUTCOMES:
change from baseline in the IBDQ at Week 8. | 0-8 weeks
Changes from baseline in fecal calprotectin over time | 0-8 weeks
Changes from baseline in serum high-sensitivity C-reactive protein (hsCRP) over time | 0-8 weeks

IPD SHARING:
Plan to Share IPD: No